CLINICAL TRIAL: NCT03848364
Title: Hip Hop Stroke: Statewide Dissemination of a School-based Public Stroke Education Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Olajide Williams, Associate Professor of Neurology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAQ6052; 2R01NS067443-06 (NIH)
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: Stroke; Education; Hip Hop Stroke; Community; Nutrition; Schools; Stroke Centers
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Stroke Centers who agree to participate will designate a Stroke coordinator who will recruit at least 2 schools from their area with 4th and/or 5th grades. Coordinators will receive a customizable electronic training package to introduce content, and recruit strategies to engage schools. They will in turn coordinate with School Champions (school designated member), who will receive program training, to implement the program. School Champion will be responsible for the distribution of Opt-Out consent forms, scheduling programming (including computer use), and coordinating with the Stroke Champion and research staff. Regarding maintenance, Stroke Coordinators and School Champions will complete and exit survey, and to promote annual implementation in recruited schools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hip Hop Stroke 2.0 intervention group (Experimental): Students in 4th and 5th grade will receive the intervention, Hip Hop Stroke 2.0, disseminated and implemented by local Stroke Centers - uses a framework of Child-Mediated Health Communication to make children "stroke literate" and then empower these stroke literate students with the tools required to successfully communicate actionable stroke knowledge (recognition of stroke symptoms and the urgency of calling 911) to their parents and grandparents at home.
  Interventions: Behavioral: Hip Hop Stroke 2.0

INTERVENTIONS:
Behavioral: Hip Hop Stroke 2.0 — HHS2.0 is an innovative, multimedia program, a brief 3-hour (1hr/day for 3 days), school-based intervention designed to educate at-risk populations concerning stroke symptoms and calling 911 immediately in the event they occur (stroke literacy). HHS2.0 is accessed and delivered via a web link online as self-administered, interactive modules that target 4th and 5th grade children in the school system (ages 9-11) using narrative cartoons and multimedia games.
  Other Names: HHS2.0

SUMMARY:
This study aims to disseminate Hip Hop Stroke 2.0 (HHS2.0) to a more heterogeneous (urban, suburban, and rural population) via NYS Stroke Centers through a partnership with the New York State Department of Health (NYSDOH) Stroke Designation Program. This digital program is a second part to an original Hip Hop Stroke program where study showed effectiveness at communicating stroke awareness. In this study, the investigator proposes to intervene in school classrooms with the Hip Hop Stroke 2.0 (HHS2.0) digital program, geared towards children aged 9 to 11 years.

Primary Aims:

Aim 1: To identify contextual factors, such as barriers and facilitators, that influence uptake of the HHS program in a new, heterogeneous sample at the Stroke Center and local school levels.

Hypothesis 1: Contextual factors at the Stroke Center and local school levels will lead to differential uptake of HHS.

Aim 2: To determine whether Stroke Center implementation of the HHS program leads to increased stroke literacy of local students by cross-validating outcomes with the results of our Randomized Clinical Trial.

Hypothesis 2: Stroke Center implementation will lead to increased stroke literacy of local students.

Secondary Aims:

Aim 3: To assess the determinants of high performance implementation and effectiveness under real world practice conditions.

Aim 4: To evaluate the costs associated with HHS program implementation.

DETAILED DESCRIPTION:
Despite effective Acute Stroke Treatment, fewer than 10% of patients in the United States receive them. The largest barrier to this treatment are pre-hospital delays which include limited to no, knowledge of stroke signs and symptoms and the intent seek care. While there is abundance of stroke education materials available, studies continue to reveal severe deficiencies in stroke literacy (knowledge of symptoms, urgent action, and prevention measures).

A mere 7% of ischemic stroke events in the US receive thrombolysis (t-PA) therapy1 due to delayed hospital arrival, most often related to the failure to recognize stroke symptoms and to call 911 immediately. Efforts to improve the public's stroke literacy have been driven by mass media stroke education campaigns that include public service announcements and print advertising. However, these efforts have failed to have an effect on 911 use (the major determinant of early hospital arrival) beyond the funding period for the specific media campaign. Stroke Centers may represent more sustainable channels for public stroke education initiatives promoting the use of ambulance services.

State Departments of Health and the Joint Commission regulate Stroke Center hospitals through an accreditation process that requires the fulfillment of certain stroke care measures. Notably, one of these regulatory requirements is community stroke education by the hospital; however, these are underdeveloped, and lack guidelines and evaluation metrics. Consequently, stroke education efforts by Stroke Centers are often poorly delivered and do not use evidence-based approaches.

The program helps schools fulfill NYS health education requirements through its primordial prevention modules. Children are also taught to teach stroke information to their parents/caregivers. HHS2.0 has shown to be effective in the real world setting through several studies, including an Randomized Clinical Trial (RCT) involving more than 3,000 predominantly Black and Hispanic urban school children aged 9-11 years. These studies found that children can and will: (1) learn how to recognize stroke, including self-efficacy for calling 911 when they witness stroke, and retain this knowledge for at least 15 months, (2) communicate stroke literacy successfully to their parents and grandparents who retain this knowledge for at least 3 months, and (3) actually call 911 when they witness stroke symptoms occurring in their homes or community.

This project is an outgrowth of our previously funded RCT (R01NS067443), in which we developed and established the effectiveness of a novel intervention to teach economically challenged minority residents of New York City to recognize stroke symptoms and know the correct response - call 911 (stroke literacy).

ELIGIBILITY:
Inclusion Criteria:

* Schools located in the 47 hospital (stroke center) geographic catchment areas
* Schools with 4th and/or 5th grade classes and have ascertained the following: student bodies have at least 50 students in each of these grades, diverse socio-demographic NYS communities, and computer resources / internet access required for the implementation of the HHS program.

Exclusion Criteria:

* Special education school with a student body comprised of those with learning disabilities.

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1706 (Actual)
Dates: Start 2015-12-17 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Stroke Literacy Score | Baseline, at least 3 days from baseline
  The Investigator will assess stroke literacy among 4th and 5th grade students with the validated Stroke Literacy Action Measure using a pre-post- test design. Literacy will be determined by percentage of questions answered correctly. The greater percentage correct indicates a better outcome.

SECONDARY OUTCOMES:
Average number of barriers influencing program uptake | Baseline, at least 1 year from baseline
  The Investigator will find the average rate of factors influencing program update through the use of the Consolidated Framework for Implementation (CFIR). The CFIR will be measured by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework to evaluate these averages.
Average number of facilitators influencing program uptake | Baseline, at least 1 year from baseline
  The Investigator will find the average rate of factors influencing program update through the use of the Consolidated Framework for Implementation (CFIR). The CFIR will be measured by the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework to evaluate these averages.
Average number of determinants yielding high performance implementation and effectiveness | Baseline, up to 2 years
  Using data from Aim 1 and Aim 2, the Investigator will analyze contextual data from each Stroke Center in relation to the data generated from RE-AIM variables. The Investigator will assess the average number of factors/elements influencing the adoption, implementation, and maintenance of the intervention at the Stroke Center and the local school level
Average total cost associated with program implementation | Baseline, up to 2 years
  The Investigator will conduct cost analyses from two complementary perspectives: 1) implementing agencies (primary cost analysis) and 2) society as a whole (secondary cost analysis). The Investigator will first estimate costs, and variations therein, based on the experience of participating Stroke Centers and schools (implementing agencies). The Investigator will develop estimates of the total cost of the HHS program, its key components and activities, and costs per participant using the resource cost method and look at the average totals.

CONTACTS AND LOCATIONS:
Overall Officials: Olajide Williams, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No